CLINICAL TRIAL: NCT02188758
Title: Do Changes in Serum Hepcidin-25 Concentration Predict Cystic Fibrosis Pulmonary Exacerbation (CFPE) Treatment Responses?
Brief Title: Biomarkers of Iron Homeostasis and Responses to Cystic Fibrosis Pulmonary Exacerbation (CFPE) Treatment
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Principal Investigator, Alex H. Gifford, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: D14136; KL2TR001088 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: iron; hepcidin-25; pulmonary exacerbation; interleukin-6
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA and RNA will be isolated from sputum samples and stored for future analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults - CFPE Treatment: Other: CF Pulmonary Exacerbation (CFPE) Treatment
  Interventions: Other: Adults - CFPE Treatment

INTERVENTIONS:
Other: Adults - CFPE Treatment — Hospitalization for comprehensive treatment of CF pulmonary exacerbation, including intravenous (IV) antibiotics, nutritional assessment and support, airway clearance of mucus, use of inhaled mucolytic agents and bronchodilators, glycemic control with insulin, and psychosocial support.

SUMMARY:
The goal of this study is to identify chemical compounds in the blood and sputum (i.e., biomarkers) that are associated with objective measurements of health status in patients with cystic fibrosis (CF). This study builds upon observations that blood levels of hepcidin-25, a protein that regulates how the body uses and stores iron, vary during CF pulmonary exacerbation (CFPE).

ELIGIBILITY:
Inclusion Criteria (required at screening visit):

* Diagnosis of CF confirmed by history of positive chloride sweat test and/or CFTR mutation analysis;
* History of consistent sputum production on most occasions;
* FEV1% greater than or equal to 75% of best measurement in previous 6 months;
* 1 or more hospitalizations for CFPE treatment with intravenous antibiotics within the previous year;
* Absence of CFPE (i.e., Akron Pulmonary Exacerbation Score <5);
* Not admitted to hospital within the previous 3 weeks;
* Body weight greater than or equal to 75% of best measurement in previous 6 months;
* Provision of signed informed-consent to study protocol;
* 18<Age>65

Exclusion Criteria:

* Women who are pregnant or lactating;
* Subject does not meet Inclusion criteria;
* Recent and/or persistent visible blood in sputum (hemoptysis);
* Rescue use of oral antibiotics within the previous 3 weeks, defined as antibiotic use for health deterioration rather than chronic suppression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater than
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Hepcidin-25 Concentration After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  The primary endpoint of this study is the characterization of 3 groups (i.e., "low," "intermediate," and "high") of serum hepcidin-25 responders to CFPE treatment. Response will be defined as the ratio of post- to pre-treatment serum hepcidin-25 concentration for each subject.

SECONDARY OUTCOMES:
Change in Percent-Predicted Forced Expiratory Volume in One Second (FEV1%) After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for FEV1% for each subject.
Change in Body Mass Index (BMI) After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for BMI for each subject.
Change in CFRSD-CRISS Score After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  CFRSD-CRISS is a patient-reported outcome (PRO) instrument developed by the Seattle Quality of Life Group at the University of Washington and used herein under license to evaluate the severity of symptoms of CF in adults and adolescents (≥12 years) with a chronic respiratory infection. Symptoms assessed in the CFRSD-CRISS are: difficulty breathing, cough, cough up mucus, chest tightness, wheeze, feeling feverish, tired, and chills/sweats. The 8 items quantify symptom severity for the previous 24 hours to capture the magnitude of symptoms in stable CF, during medically treated CF exacerbations, and during recovery from an exacerbation. We will determine the within-subject differences in CFRSD-CRISS score associated with CFPE treatment.
Change in Serum Iron After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum iron concentration for each subject.
Change in Serum Interleukin-6 (IL-6) Concentration After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum interleukin-6 (IL-6) concentration for each subject.
Change in Sputum Iron Content After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for sputum iron content for each subject.
Change in Serum EPO Concentration After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum erythropoietin (EPO) for each subject.
Change in Transferrin Saturation After Hospitalization for CF Pulmonary Exacerbation Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for transferrin saturation for each subject.
Change in Serum TREM-1 Concentration After Hospitalization for CF Pulmonary Exacerbation Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum triggering receptor expressed on myeloid cells-1 (TREM-1) for each subject.
Change in Serum sIL-6R Concentration After Hospitalization for CF Pulmonary Exacerbation Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum soluble IL-6 receptor (sIL-6R) concentration for each subject.
Change in Hemoglobin Concentration After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for serum hemoglobin concentration for each subject.

OTHER OUTCOMES:
Change in Sputum SDI After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratio for Simpson Diversity Index (SDI) for each subject.
Change in Sputum Pseudomonas aeruginosa Gene Expression After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratios for selected Pseudomonas aeruginosa mRNA transcript levels.
Change in Peripheral Blood Mononuclear Cell (PBMC) Gene Expression After Hospitalization for CF Pulmonary Exacerbation (CFPE) Treatment | Duration of hospitalization, an expected average of 12 days
  Post- to pre-treatment ratios for selected mRNA transcript levels.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Maine Medical Center, South Portland, Maine
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] Gifford AH. What is hepcidin telling us about the natural history of cystic fibrosis? J Cyst Fibros. 2015 Jan;14(1):155-7. doi: 10.1016/j.jcf.2014.03.012. Epub 2014 Apr 30. No abstract available. PMID 24795218
- [Background] Gifford AH, Alexandru DM, Li Z, Dorman DB, Moulton LA, Price KE, Hampton TH, Sogin ML, Zuckerman JB, Parker HW, Stanton BA, O'Toole GA. Iron supplementation does not worsen respiratory health or alter the sputum microbiome in cystic fibrosis. J Cyst Fibros. 2014 May;13(3):311-8. doi: 10.1016/j.jcf.2013.11.004. Epub 2013 Dec 13. PMID 24332997
- [Background] Gifford AH. Hemoglobin </= 12.9 g/dl predicts risk of antibiotic treatment in cystic fibrosis. J Cyst Fibros. 2014 Jan;13(1):114-5. doi: 10.1016/j.jcf.2013.06.007. Epub 2013 Jul 16. No abstract available. PMID 23867071
- [Background] Gifford AH, Moulton LA, Dorman DB, Olbina G, Westerman M, Parker HW, Stanton BA, O'Toole GA. Iron homeostasis during cystic fibrosis pulmonary exacerbation. Clin Transl Sci. 2012 Aug;5(4):368-73. doi: 10.1111/j.1752-8062.2012.00417.x. Epub 2012 Jun 1. PMID 22883617
- [Background] Gifford AH, Miller SD, Jackson BP, Hampton TH, O'Toole GA, Stanton BA, Parker HW. Iron and CF-related anemia: expanding clinical and biochemical relationships. Pediatr Pulmonol. 2011 Feb;46(2):160-5. doi: 10.1002/ppul.21335. Epub 2010 Oct 20. PMID 20963784